CLINICAL TRIAL: NCT02329496
Title: REPRISE NGDS: REpositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of LotuS™ ValvE With the Next Generation Delivery System
Brief Title: REPRISE Next Generation Delivery System
Acronym: NGDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2332
Record Dates: First submitted 2014-11-19; First posted 2014-12-31 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lotus Valve and LOTUS Edge Valve System (Experimental): Transcatheter aortic valve replacement (TAVR) with Lotus Valve System with the Next Generation Delivery System and LOTUS Edge Valve System
  Interventions: Device: Lotus Valve and LOTUS Edge Valve System

INTERVENTIONS:
Device: Lotus Valve and LOTUS Edge Valve System — Transcatheter aortic valve replacement (TAVR) with the Lotus Valve System with the Next Generation Delivery System and LOTUS Edge Valve System, with either the Lotus Introducer or iSleeve Introducer Sets

SUMMARY:
To confirm the acute performance and safety of the Lotus™ Valve with the Next Generation Delivery System for transcatheter aortic valve replacement (TAVR) in symptomatic patients with severe calcific aortic stenosis who are considered high risk for surgical valve replacement.

DETAILED DESCRIPTION:
This clinical study is a prospective single-arm study designed to demonstrate that the acute performance and safety of the LOTUS Edge Valve System when used with the iSleeve Introducer Set or current Lotus Introducer Set are consistent with the results of the Lotus Valve System used in the REPRISE II study, when delivered and deployed in symptomatic subjects who have severe calcific aortic valve stenosis and who are at high risk for surgical aortic valve replacement (SAVR).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥70 years of age
2. Subject has documented calcific native aortic valve stenosis with an initial aortic valve area (AVA) of ≤1.0 cm2 (or AVA index of ≤0.6 cm2/m2) and either a mean pressure gradient ≥40 mm Hg or a jet velocity ≥4 m/s, as measured by echocardiography.
3. Subject has a documented aortic annulus size between ≥20 and ≤27.5 mm based on pre-procedure diagnostic imaging
4. Subject has symptomatic aortic valve stenosis with NYHA Functional Class ≥ II.
5. Subject is considered high risk for surgical valve replacement based on at least one of the following:

   * Society of Thoracic Surgeons (STS) score ≥8%, and/or
   * Agreement by the heart team (which must include an in-person evaluation by an experienced cardiac surgeon) that subject is at high operative risk of serious morbidity or mortality with surgical valve replacement.
6. Heart team (which must include an experienced cardiac surgeon) assessment that the subject is likely to benefit from valve replacement
7. Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.
8. Subject, family member and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion Criteria:

1. Subject has a congenital unicuspid or bicuspid aortic valve.
2. Subject with an acute myocardial infarction within 30 days of the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of creatine kinase-myoglobin band (CK-MB) elevation and/or troponin level elevation).
3. Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months, or has any permanent neurologic defect prior to study enrollment.
4. Subject is on dialysis or has serum creatinine level >3.0 mg/dL or 265 µml/L.
5. Subject has a pre-existing prosthetic heart valve (aortic or mitral) or a prosthetic ring in any position.
6. Subject has ≥3+ mitral regurgitation, ≥3+ aortic regurgitation or ≥3+ tricuspid regurgitation (i.e., subject cannot have more than moderate mitral, aortic or tricuspid regurgitation).
7. Subject has a need for emergency surgery for any reason.
8. Subject has a history of endocarditis within 12 months of index procedure or evidence of an active systemic infection or sepsis.
9. Subject has echocardiographic evidence of intra-cardiac mass, thrombus or vegetation.
10. Subject has Hgb <9 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
11. Subject is receiving chronic (≥72 hours) anticoagulation therapy (warfarin), and cannot tolerate concomitant therapy with aspirin or clopidogrel (subjects who require chronic anticoagulation must additionally be able to be treated with either aspirin or clopidogrel).*
12. Subject has active peptic ulcer disease or gastrointestinal bleed within the past 3 months, other bleeding diathesis or coagulopathy or will refuse transfusions.
13. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all thienopyridines, heparin, nickel, titanium, or polyurethanes.
14. Subject has a life expectancy of less than 12 months due to non-cardiac, co-morbid conditions based on the assessment of the investigator at the time of enrollment.
15. Subject has hypertrophic obstructive cardiomyopathy.
16. Subject has any therapeutic invasive cardiac procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty and pacemaker implantation which are allowed).
17. Subject has untreated coronary artery disease, which in the opinion of the treating physician, is clinically significant and requires revascularization.
18. Subject has documented left ventricular ejection fraction <30%.
19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
20. Subject has severe peripheral vascular disease (including aneurysm defined as maximal luminal diameter >5 cm or with documented presence of thrombus, marked tortuosity, narrowing of the abdominal aorta, severe unfolding of the thoracic aorta or thick [>5 mm] protruding or ulcerated atheroma in the aortic arch) or symptomatic carotid or vertebral disease.
21. Femoral artery lumen of <6.0 mm for subjects requiring 23 mm valve size or <6.5 mm for subjects requiring 27 mm valve size, or severe iliofemoral tortuosity or calcification that would prevent safe placement of the introducer sheath.
22. Current problems with substance abuse (e.g., alcohol, etc.).
23. Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
24. Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2016-10-06 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Technical Success | Immediately post-procedure (patient discharged from operative room)
  Defined as successful vascular access, delivery, and deployment of the Lotus Valve; successful retrieval with the Lotus Next Generation delivery system; and correct positioning of a single Lotus Valve in the proper anatomical location (reported as percent of subjects implanted with a Lotus Valve). Reported as percent of subjects.

SECONDARY OUTCOMES:
Successful repositioning of the study valve if repositioning is attempted | Immediately post-procedure (patient discharged from operative room)
  Reported as percent of subjects
Successful retrieval of the study valve if retrieval is attempted | Immediately post-procedure (patient discharged from operative room)
  Reported as percent of subjects
Severe or moderate paravalvular aortic regurgitation as measured by echocardiography and assessed by an independent core laboratory | At discharge from hospital or at 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Mild, trace/trivial, or no paravalvular aortic regurgitation as measured by echocardiography and assessed by an independent core laboratory | At discharge from hospital or at 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Mean aortic valve pressure gradient as measured by echocardiography and assessed by an independent core laboratory | At discharge from hospital or at 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as mean ± standard deviation; mmHg
Effective orifice area as measured by echocardiography and assessed by an independent core laboratory | At discharge from hospital or at 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as mean ± standard deviation; cm2
Peak aortic valve pressure gradient as measured by echocardiography and assessed by an independent core laboratory | At discharge from hospital or at 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as mean ± standard deviation; mmHg
Peak aortic velocity as measured by echocardiography and assessed by an independent core laboratory | At discharge from hospital or at 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as mean ± standard deviation; m/sec
Mortality: all-cause, cardiovascular, and non-cardiovascular | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Stroke: disabling and non-disabling | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Myocardial infarction (MI): periprocedural (≤72 hours post index procedure) and spontaneous (>72 hours post index procedure) | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Bleeding: life-threatening (or disabling) and major | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Acute kidney injury based on the Acute Kidney Injury Network (AKIN) System Stage 3 (including renal replacement therapy) or Stage 2 | ≤7 days post index procedure
  Reported as percent of subjects
Major vascular complications major | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Repeat procedure for valve-related dysfunction (surgical or interventional therapy) | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Hospitalization for valve-related symptoms or worsening congestive heart failure (NYHA class III or IV) | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
New permanent pacemaker implantation resulting from new or worsened conduction disturbances | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
New onset of atrial fibrillation or atrial flutter | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Coronary obstruction | ≤72 hours post index procedure
  Reported as percent of subjects
Ventricular septal perforation | ≤72 hours post index procedure
  Reported as percent of subjects
Mitral apparatus damage | ≤72 hours post index procedure
  Reported as percent of subjects
Cardiac tamponade | ≤72 hours post index procedure
  Reported as percent of subjects
Prosthetic aortic valve malpositioning, including valve migration, valve embolization, or ectopic valve deployment | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Transcatheter aortic valve (TAV)-in-TAV deployment | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Prosthetic aortic valve thrombosis | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Prosthetic aortic valve endocarditis | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Neurological status per modified Rankin Scale score | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Neurological status per National Institutes of Health Stroke Scale | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects
Functional Improvement from baseline per NYHA functional classification | At discharge from hospital or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 12 months post procedure
  Reported as percent of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gooley, MD, Principal Investigator — Monash
Locations (2):
- Australia (2):
  - Prince Charles Hospital, Chermside, Queensland
  - Monash Heart, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No